CLINICAL TRIAL: NCT03783962
Title: Examining Cooking as a Health Behavior
Acronym: iChef
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Jean R. Harvey, PhD, RD, Chairperson, Professor, Associate Dean, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBSS 19-0131
Record Dates: First submitted 2018-12-05; First posted 2018-12-21 (Actual); Results first posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Obesity
Keywords: behavioral weight loss intervention, obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The Behavioral Weight Loss Program: Investigators have developed and implemented a theory-based group-delivered behavioral weight control program in two previous studies that incorporates the elements of current thinking and empirical data on successful weight loss programs, including restricted calorie intake and increased physical activity. In addition to attending weekly classes, participants will track their food intake, exercise, and weight. Participants will share online tracking diaries with the group facilitator who will offer individualized feedback on progress.
  The Cooking Program Active Intervention. Twelve cooking classes will be run every other week after the in-person weight loss meetings.
  Demonstrations. The demonstration condition will serve as an "attention only" control. All participants will have an opportunity to sample the prepared food at the end of class. The demonstrations will be led by the same chef as the active intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Intervention - Cooking (Experimental): Twelve cooking classes will be run every other week after the in-person weight loss meetings. These lessons will be patterned after Dr. Amy Trubek's cooking pedagogy and will be tailored for individuals specifically interested in weight loss. Classes will begin with a brief lecture on the day's topic, followed by a laboratory session. Participants work in teams of two in the Nutrition and Food Sciences (NFS) foods lab to actively practice skills and cook a meal. Subjects will receive recipes and information sheets that cover pantry supplies, grocery lists, knife skills and cooking equipment. Classes will be taught by a chef trained in the pedagogy by Dr. Trubek and participants will have the opportunity to sample the food they prepared at the end of class.
  Interventions: Behavioral: Active Intervention - Cooking
- Demonstrations - Cooking (Active Comparator): The demonstration condition will serve as an "attention only" control. Previous research suggests that demonstrations of cooking have little to no impact on cooking behavior, therefore, cooking demonstrations can be used to "even out" the time and attention devoted to the active cooking participants without introducing bias into the study design. Subjects in the demonstration condition will also begin with a brief lecture on the day's lesson followed by a cooking demonstration that covers the same topics as the active intervention group. All participants will receive the same printed information and also have an opportunity to sample the prepared food at the end of class. The demonstrations will be led by the same chef as the active intervention group.
  Interventions: Behavioral: Demonstrations - Cooking

INTERVENTIONS:
Behavioral: Active Intervention - Cooking — Key behavioral strategies to facilitate making sustained changes in dietary habits and activity patterns are introduced, promoted and reinforced throughout the program. In-person sessions facilitated by an interventionist provide the group meetings. The program provides 24 weekly facilitated group sessions over 6 months. In addition to attending weekly classes, participants will track food intake, exercise, and weight. Participants will share online tracking diaries with the group facilitator who will offer individualized feedback on individual progress.
  Twelve cooking classes will be run every other week after the in-person weight loss meetings.
  Arms: Active Intervention - Cooking
Behavioral: Demonstrations - Cooking — The Demonstrations group will receive the exact same behavioral weight loss intervention as the cooking group. The only difference is that this group will attend cooking demonstrations as opposed to actively cooking.
  Arms: Demonstrations - Cooking

SUMMARY:
The proposed pilot study will examine cooking as an intervention target for weight control in overweight adults. The study will also examine whether interventions designed to promote cooking at home can increase participants' sense of food agency, and overcome common barriers to cooking at home such as time scarcity and budget constrictions. The study will utilize a cooking pedagogy designed to not just teach participants the basics of cooking different foods, but how to be efficient, mindful cooks. If cooking class participation positively impacts diet and health outcomes, it will bolster the case for promoting cooking at home as a health behavior for multiple populations.

DETAILED DESCRIPTION:
A two arm randomized control trial will examine whether the addition of an active cooking lesson versus a passive observed lesson to a behavioral weight loss intervention results in significantly greater weight loss. Additionally, the study will examine whether interventions designed to promote cooking at home can increase participants' sense of food agency, and overcome common barriers to cooking at home such as time scarcity and budget constrictions.

Overweight and obese but otherwise healthy participants (n=64) will be recruited. Recruitment and study initiation will occur in two waves. Wave 1 aims to recruit 32 individuals who will then be randomized to 1) a 24 week, 24 session group behavioral weight loss intervention with 12 bi-weekly cooking lessons; or, 2) the same 24 week, 24 session group behavioral weight loss intervention with 12 bi-weekly cooking demonstrations. Both groups get the same intervention and the same counselor delivered intervention elements; the presence of active cooking lessons vs. passive observed cooking demonstrations is the only difference between conditions. Assessments will be conducted at 0, 3 and 6 months. Wave 2 (n=32) will follow the same process as Wave 1 approximately two months after Wave 1 is initiated.

ELIGIBILITY:
Inclusion Criteria:

* only individuals who are cooking (from scratch) no more than 3 meals at home per week will be eligible.
* must have a computer or smart device with internet access (at home or work) in order to track their diet and exercise behaviors,
* potential participants will be required to demonstrate some ability to comply with study intervention procedures to be eligible (specifically, they must complete an online dietary self-monitoring diary for 3 days)
* must be at least 18 years old and have a BMI between 25-50 kg/m2
* must agree to be randomized to either study arm and available for both scheduled meeting times in person on the University of Vermont campus

Exclusion Criteria:

* pregnant or planning to become pregnant in the next 6 months or lactating
* physical conditions that would preclude exercise
* medication affecting weight loss
* currently enrolled in another weight loss program
* currently cooking more than 3 meals from scratch at home per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean R Harvey, PhD, RD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Intervention - Cooking: Twelve cooking classes will be run every other week after the in-person weight loss meetings. These lessons will be patterned after Dr. Amy Trubek's cooking pedagogy and will be tailored for individuals specifically interested in weight loss. Classes will begin with a brief lecture on the day's topic, followed by a laboratory session. Participants work in teams of two in the NFS foods lab to actively practice skills and cook a meal. Subjects will receive recipes and information sheets that cover pantry supplies, grocery lists, knife skills and cooking equipment. Classes will be taught by a chef trained in the pedagogy by Dr. Trubek and participants will have the opportunity to sample the food they prepared at the end of class.
  Active Intervention - Cooking: Key behavioral strategies to facilitate making sustained changes in dietary habits and activity patterns are introduced, promoted and reinforced throughout the program. In-person sessions facilitated by an interventionist provide the group meetings. The program provides 24 weekly facilitated group sessions over 6 months. In addition to attending weekly classes, participants will track food intake, exercise, and weight. Participants will share online tracking diaries with the group facilitator who will offer individualized feedback on individual progress.
  Twelve cooking classes will be run every other week after the in-person weight loss meetings.
Period: Overall Study
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Started | 28 | 28
Completed | 25 | 21
Not Completed | 3 | 7
Not completed — Lost to Follow-up | 3 | 6
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Intervention - Cooking: Twelve cooking classes will be run every other week after the in-person weight loss meetings. These lessons will be patterned after Dr. Amy Trubek's cooking pedagogy and will be tailored for individuals specifically interested in weight loss. Classes will begin with a brief lecture on the day's topic, followed by a laboratory session. Participants work in teams of two in the University of Vermont Nutrition and Food Sciences department foods lab to actively practice skills and cook a meal. Subjects will receive recipes and information sheets that cover pantry supplies, grocery lists, knife skills and cooking equipment. Classes will be taught by a chef trained in the pedagogy by Dr. Trubek and participants will have the opportunity to sample the food they prepared at the end of class.
  Active Intervention - Cooking: Key behavioral strategies to facilitate making sustained changes in dietary habits and activity patterns are introduced, promoted and reinforced throughout the program. In-person sessions facilitated by an interventionist provide the group meetings. The program provides 24 weekly facilitated group sessions over 6 months. In addition to attending weekly classes, participants will track food intake, exercise, and weight. Participants will share online tracking diaries with the group facilitator who will offer individualized feedback on individual progress.
  Twelve cooking classes will be run every other week after the in-person weight loss meetings.
- Total: Total of all reporting groups
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 28 | 55
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (11) | 50 (11) | 53 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White or Euro-American | 28 | 24 | 52
  Middle Eastern or Arab American | 0 | 1 | 1
  Latino or Hispanic American | 0 | 1 | 1
  Other | 0 | 1 | 1
  Prefer not to answer | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56
Education [Count of Participants; unit: Participants]
  High School graduate, GED, Some college | 8 | 7 | 15
  College Degree | 10 | 15 | 25
  Graduate Degree, Professional Education | 10 | 6 | 16
Marital Status [Count of Participants; unit: Participants]
  Married | 16 | 17 | 33
  Separated | 0 | 1 | 1
  Divorced | 5 | 4 | 9
  Never Married | 6 | 6 | 12
  Widowed | 1 | 0 | 1
Employment [Count of Participants; unit: Participants]
  Employed | 23 | 26 | 49
  Retired | 2 | 1 | 3
  Disabled | 1 | 1 | 2
  Homemaker | 1 | 0 | 1
  Not currently employed | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: Weight loss from baseline at 24 weeks
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Deviation); unit: kilogram
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 27 | 23
kilogram | 7.34 (.63) | 4.49 (.67)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .003, Mixed Models Analysis

2. Primary Outcome: Change From Baseline in the Total HEI Score, as a Measure of Diet Quality Change
Description: Difference in diet quality change between groups across assessments. Measured by Healthy Eating Index scores.
  The HEI includes 13 components that capture recommendations of the 2015-2020 Dietary Guidelines for Americans. There are two groupings of components:
  1. Adequacy components are encouraged. Higher scores reflect higher intakes.
  2. Moderation components should be limited. Higher scores reflect lower intakes. A higher total HEI score reflects higher diet quality as defined by the Dietary Guidelines for Americans.
  Components are weighted equally and assigned a score of either 5 or 10. Scores as summed to determine total score. The minimum possible score is 0 and the maximum possible is 100.
  Adequacy Components:
  Total Fruits 5 Whole Fruits 5 Total vegetables 5 Greens and beans 5 Whole grains 10 Dairy 10 Total protein foods 5 Seafood and plant proteins 5 Fatty acids 10
  Moderation Components:
  Refined grains 10 Sodium 10 Added sugars 10 Saturated fats 10
Time Frame: Baseline and 24 weeks
Measure: Least Squares Mean (Standard Deviation); unit: points
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 18
points | 6.08 (2.62) | 6.23 (2.84)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .97, Mixed Models Analysis

3. Secondary Outcome: Cooking and Food Practices Change - Total Score
Description: Difference in baseline and end point Cooking and Food Provisioning Action Scale Total scores between groups.
  Structure subscale measures whether an individual thinks their cooking ability and skills are adequate. On a scale of 1-21, higher scores over time indicate improvement.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
score on a scale
  Total Score baseline | 11.25 (.37) | 10.41 (.37)
  Total Score 24 weeks | 13.34 (.4) | 13.4 (.41)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .08, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis

4. Secondary Outcome: Cooking and Food Practices Change - Structure Subscale
Description: Difference in baseline and end point Cooking and Food Provisioning Action Scale Structure subscale scores between groups.
  Structure subscale measures the ways in which external factors can either hinder or support an individual's cooking and provisioning actions. On a scale of 1-7, higher scores over time indicate improvement.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
score on a scale
  Structure baseline | 3.20 (.19) | 2.74 (.19)
  Structure 24 weeks | 3.37 (.20) | 3.32 (.21)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .18, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p = .40, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p = .01, Mixed Models Analysis

5. Secondary Outcome: Cooking and Food Practices Change - Attitude Subscale
Description: Difference in baseline and end point Cooking and Food Provisioning Action Scale Attitude subscale scores between groups.
  Structure subscale measures an individual's affective stance towards food, cooking and provisioning in different areas. On a scale of 1-7, higher scores over time indicate improvement.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
score on a scale
  Attitude baseline | 4.45 (.17) | 4.32 (.17)
  Attitude 24 weeks | 5.31 (.18) | 5.37 (.19)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .40, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis

6. Secondary Outcome: Cooking and Food Practices Change - Self Efficacy Subscale
Description: Difference in baseline and end point Cooking and Food Provisioning Action Scale Self Efficacy subscale scores between groups.
  Structure subscale measures whether an individual thinks their cooking ability and skills are adequate. On a scale of 1-7, higher scores over time indicate improvement.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
score on a scale
  Self Efficacy baseline | 3.59 (.15) | 3.35 (.15)
  Self Efficacy 24 weeks | 4.65 (.17) | 4.70 (.18)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .25, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis

7. Secondary Outcome: Cooking Frequency Change - Breakfast
Description: Breakfast cooking frequency was assessed at baseline and 24 weeks using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: 24 weeks
Measure: Mean (Standard Error); unit: meals cooked
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
meals cooked
  Breakfast baseline | 2.46 (.37) | 1.54 (.37)
  Breakfast 24 weeks | 2.82 (.41) | 1.07 (.34)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .26, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p = .41, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p = .02, Mixed Models Analysis

8. Secondary Outcome: Cooking Frequency Change - Lunch
Description: Lunch cooking frequency was assessed at baseline and 24 weeks using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: meals cooked
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
meals cooked
  Lunch baseline | 1.07 (.34) | 1.07 (.34)
  Lunch 24 weeks | 2.17 (.38) | 3.58 (.40)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .03, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p = .02, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p < .001, Mixed Models Analysis

9. Secondary Outcome: Cooking Frequency Change - Dinner
Description: Dinner cooking frequency was assessed at baseline and 24 weeks using the cooking frequency subscale from the Cooking Perceptions/Attitudes/Confidence/Behaviors Survey. The scores range from a minimum of 0 to a maximum of 7 meals cooked during a one week period.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: meals cooked
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 23 | 19
meals cooked
  Dinner baseline | 2.57 (.33) | 3.25 (.33)
  Dinner 24 weeks | 3.37 (.36) | 4.38 (.39)
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .58, Mixed Models Analysis
Statistical Analysis 2: Comparison: Active Intervention - Cooking; Test type: Superiority; p = .05, Mixed Models Analysis
Statistical Analysis 3: Comparison: Demonstrations - Cooking; Test type: Superiority; p = .01, Mixed Models Analysis

10. Secondary Outcome: Treatment Engagement- Attendance
Description: Percent (of 24 possible) classes attended will be calculated to determine treatment engagement
Time Frame: 24 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of classes attended
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 28 | 28
percentage of classes attended | 83 [77 to 87] | 69 [29 to 83]
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = .009, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Treatment Engagement- Food Journaling Compliance
Description: Percent of weekly food journals at least partially completed (an entry made during a seven day period) will be calculated to determine treatment engagement
Time Frame: Baseline to six months
Measure: Median (Inter-Quartile Range); unit: percentage of complete food journals
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
Number analyzed (Participants) | 27 | 23
percentage of complete food journals | 95.92 [72.00 to 100] | 87.75 [35.42 to 98]
Statistical Analysis 1: Comparison: Active Intervention - Cooking vs Demonstrations - Cooking; Test type: Superiority; p = 0.12, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Baseline to 6 months
Arm/Group | Active Intervention - Cooking | Demonstrations - Cooking
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03783962/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03783962/ICF_000.pdf